CLINICAL TRIAL: NCT05031169
Title: Evaluation of Surgical Management of Interdental Papilla Recession With Advanced Platelet Rich Fibrin Compared to Subepthelial Connective Tissue Graft. A Randomized Controlled Trial
Brief Title: Surgical Management of Interdental Papilla Recession With Advanced Platelet Rich Fibrin or Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sanabel Osama Omran Barakat, Ph d candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER 331
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Recession
Keywords: interdental papilla reconstriction

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-PRF (Experimental): Surgical treatment A-PRF membrane
  Interventions: Procedure: interdental papilla surgical reconstructiion
- SCTG (Active Comparator): Surgical treatment with SCTG
  Interventions: Procedure: interdental papilla surgical reconstructiion

INTERVENTIONS:
Procedure: interdental papilla surgical reconstructiion — Surgical treatment of receding interdentalpapillae

SUMMARY:
deficient interdental papillae witt be surgically reconstructed. in one group, connective tissue graft (SCTG) will be used for papillae augmentation, while in the other group, advanced platelet rich fibrin (A-PRF). the height of the papillae will be measured preoperatively as well as post operatively at 3, 6 ,9 and 12 months.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of A-PRF membrane to SCTG when used as grafting material with the Han and Takei's approach to reconstruct receding interdental papilla and assess deference in papilla height between the study groups.

The clinical parameters that will be evaluated are:

* Papilla height (PH)
* Clinical attachment level (CAL)
* Probing depth (PD)
* Post-operative patients' satisfaction about the esthetic outcome
* Post-operative pain level among patients

Study settings:

This study will be conducted in the postgraduate periodontology clinics in the faculty of dentistry, Cairo University. The participants will be selected from the outpatient clinic of the department.

interventionsa:

The first visit:

* Eligible participants will be interviewed to report medical and dental histories.
* The participants will receive full mouth dental and periodontal examination.
* Initial periodontal treatment (supragingival scaling and sub gingival debridement) as indicated.
* Patients will be given oral hygiene instruction on proper tooth brushing and flossing.
* They will be advised to use chlorhexidine mouth wash 0.12% twice daily for 2 weeks.

Second visit:

After 4-6 weeks of initial therapy, patients will be re-examined, and the baseline clinical parameters will be recorded as follows:

* Full mouth plaque index and gingival index.
* Site specific plaque index and gingival index.
* Type of Papilla deficiency (classification).
* Papilla height
* Clinical attachment level
* Probing depth

The patients then will be randomly allocated to one of the study groups.

Test group:

Deficient papillae in this group will be treated surgically and A-PRF membrane will be used as a grafting material.

Preparation of A-PRF:

A-PRF preparation protocol will be as described by (Clark et al. 2018):

A blood sample of 10 ml will be obtained from the patient and immediately centrifuged at 1300 rpm for 8 minutes.

Control group:

In this group, papilla recession will be treated surgically and the SCTG will be used as a grafting material.

sample size calculation was based on a previous study. fourteen experimental subjects and 14 control subjects are required to be able to reject the null hypothesis that the population means of the experimental and the control groups are equal with probability (power) 0.8. The type I error probability associated with this test of this null hypothesis is 0.05.

To compensate for anticipated missing data during follow up, this number is increased to 16 per group.

Recruitment

* Patients will be selected from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Oral and Dental Medicine-Cairo University
* Screening of patients will continue until the target sample is achieved.

Allocation

Randomization:

Patients will be randomly assigned to either test or control group using computer generated randomization (www.randomizer.org) which will be performed by the supervisor. The patients will be allocated to either test or control group.

Allocation concealment mechanism:

The two groups will be equally prepared for both surgical procedures. Then the decision of which group will receive papilla treatment with A-PRF (test) and which will receive papilla treatment with SCTG (control) will be taken according to the randomized numbers placed in opaque sealed envelopes. The number will be picked by the supervisor.

Implementation:

• All patients who provide an informed consent for participation as well as fulfill the inclusion criteria will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy adults older than 18 years of age and presenting at least one deficient papilla with papilla presence index 2 or 3
* Have Interproximal CAL ≤ 3 mm
* Have probing depth ≤ 3mm
* Distance between the alveolar bone crest and contact point is less than 7mm.

Exclusion Criteria:

* Smoking.
* Pregnancy and lactation.
* Carious and non-carious cervical lesion in the involved teeth around the papilla.
* Restoration in teeth around the papilla (filling, crown, bridge, facings, clasp of a partial denture).
* Open contacts and non-vital teeth
* Poor oral hygiene with plaque index > 20 %.
* Tooth mobility
* History of medication in the previous 3 months
* History of periodontal surgery in the site to be treated in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
papilla height | base line , 3, 6, 9, and 12 months
  change of papillae height will be recorded using a graduated periodontal probe (UNC 15 probe)

SECONDARY OUTCOMES:
patient satisfaction | 3 and 12 months
  patients opinion about esthetic improvement

CONTACTS AND LOCATIONS:
Overall Officials: Hani ElNahass, Ph D, Study Chair — Cairo University; Samar ElKohouly, Ph D, Principal Investigator — Cairo University; sanabel barakat, MSC, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahila E, Saravana Kumar R, Reddy VK, Pratebha B, Jananni M, Priyadharshini V. Augmentation of Interdental Papilla with Platelet-rich Fibrin. Contemp Clin Dent. 2018 Apr-Jun;9(2):213-217. doi: 10.4103/ccd.ccd_812_17. PMID 29875563
- [Background] Cardaropoli D, Re S, Corrente G, Abundo R. Reconstruction of the maxillary midline papilla following a combined orthodontic-periodontic treatment in adult periodontal patients. J Clin Periodontol. 2004 Feb;31(2):79-84. doi: 10.1111/j.0303-6979.2004.00451.x. PMID 15016030
- [Background] Augusta, Maria and Matas Hennig. 2016. "Absence of Interdental Papilla - Systematic Review of Available Therapeutic Modalities." Stomatos 22(43):31-43.
- [Background] Chaulkar PP, Mali RS, Mali AM, Lele PA, Patil PA. A comparative evaluation of papillary reconstruction by modified Beagle's technique with the Beagle's surgical technique: A clinical and radiographic study. J Indian Soc Periodontol. 2017 May-Jun;21(3):218-223. doi: 10.4103/jisp.jisp_166_17. PMID 29440789
- [Background] Clark D, Rajendran Y, Paydar S, Ho S, Cox D, Ryder M, Dollard J, Kao RT. Advanced platelet-rich fibrin and freeze-dried bone allograft for ridge preservation: A randomized controlled clinical trial. J Periodontol. 2018 Apr;89(4):379-387. doi: 10.1002/JPER.17-0466. PMID 29683498
- [Background] Eren G, Atilla G. Platelet-rich fibrin in the treatment of localized gingival recessions: a split-mouth randomized clinical trial. Clin Oral Investig. 2014 Nov;18(8):1941-8. doi: 10.1007/s00784-013-1170-5. Epub 2013 Dec 22. PMID 24362634
- [Background] Ghanaati S, Booms P, Orlowska A, Kubesch A, Lorenz J, Rutkowski J, Landes C, Sader R, Kirkpatrick C, Choukroun J. Advanced platelet-rich fibrin: a new concept for cell-based tissue engineering by means of inflammatory cells. J Oral Implantol. 2014 Dec;40(6):679-89. doi: 10.1563/aaid-joi-D-14-00138. PMID 24945603